CLINICAL TRIAL: NCT01998685
Title: Prothrombotic Factors , Angiogenic Growth Factor and Different Anaesthetic Techniques in Cancer Patients Undergoing Prostatectomy
Brief Title: Prothrombotic Factors and Anaesthesia in Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Principal Investigator, Ester Forastiere, chief, Regina Elena Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 550
Record Dates: First submitted 2013-11-13; First posted 2013-12-02 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Prostatic Cancer; Surgery
Keywords: Prostatectomy; Coagulation Factor; Balanced Anesthesia; Intravenous Anesthesia,
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Propofol; Remifentanil; Midazolam; Fentanyl; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Balanced (BAL) anaesthesia (Experimental): In the BAL group anaesthesia is induced with midazolam 0.1mg kg-1 and fentanyl 1.5 μg kg- 1 Anaesthesia is maintained with sevoflurane 2.0% , oxygen 40% and air 70% with positive pressure ventilation in a circle system, in order to achieve normocapnia.
  Interventions: Drug: Midazolam; Drug: Fentanyl; Drug: Sevoflurane
- Totally Intravenous Anesthesia (TIVA-TCI) (Active Comparator): In the TIVA-TCI group anaesthesia is induced with propofol 6 microg ml-1 and remifentanyl 0.4-1 microg kg-1 min, simultaneously administered using two separate modules of a continuous computer-assisted TCI system. Anaesthesia is maintained with propofol 4 microg ml-1 and remifentanil 0.25 microg Kg-1 min. This infusion is modified by 0.05 microg kg-1 min steps according to analgesic needs.
  Interventions: Drug: Propofol; Drug: remifentanyl

INTERVENTIONS:
Drug: Propofol
  Other Names: Diprivan
  Arms: Totally Intravenous Anesthesia (TIVA-TCI)
Drug: remifentanyl
  Other Names: Ultiva
  Arms: Totally Intravenous Anesthesia (TIVA-TCI)
Drug: Midazolam
  Arms: Balanced (BAL) anaesthesia
Drug: Fentanyl
  Other Names: Fentanest
  Arms: Balanced (BAL) anaesthesia
Drug: Sevoflurane
  Other Names: Sevorane
  Arms: Balanced (BAL) anaesthesia

SUMMARY:
This study aims to assess if different anesthetic techniques can affect coagulant factors in patients with prostate cancer undergoing elective laparoscopic radical prostatectomy (LRP).

DETAILED DESCRIPTION:
The utility of anti-thrombotic prophylaxis in cancer patients undergoing laparoscopic radical prostatectomy (LRP) is still controversial. Moreover, different anaesthetic techniques could modify coagulant factors. Thus, in this study we will be to investigate the variations of pro- and anti-coagulant and fibrinolytic factors in two established types of anaesthesia in patients with prostate cancer undergoing elective LRP.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed cancer of the prostate
* histological Gleason score evaluation.

Exclusion Criteria:

* ASA >2
* metabolic equivalent task < 4
* BMI>30
* no pre-operative pharmacological thromboprophylaxis and/or anti-coagulant therapy
* history of abnormal bleeding, or abnormal coagulant factors
* sepsis within the last 2 weeks
* previous new adjuvant treatments (chemo, hormone, and radiotherapy)
* non-steroid , anti-inflammatory and statins drugs for at least 2 wks before surgery
* venous or arterial thromboembolism within the last 3 months, peripheral venous disease
* neurological disease with extremity paresis
* chronic liver disease
* pre-operative haemoglobin concentration < 9 mg dl-1
* prolonged duration of surgery (>3 hrs)
* peri-operative blood transfusion
* not adequate material for laboratory testing

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Rate of rate of prothrombotic markers and Vascular Endothelial Growth Factor (VEGF) variation | 24 hours

SECONDARY OUTCOMES:
Free-desease survivall | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ester Forastiere, MD, Study Director — Department of Anaesthesiology, Regina Elena, National Cancer Institute, Via Elio Chianesi 53, 00144 Roma (Italy); Tel. +39 0652662942, FAX: +39 0652662993; e-mail: forastiere@ifo.it
Locations (1):
- Department of Anaesthesiology, Regina Elena, National Cancer Institute, Roma, Italy

REFERENCES:
- [Derived] Sofra M, Antenucci A, Gallucci M, Mandoj C, Papalia R, Claroni C, Monteferrante I, Torregiani G, Gianaroli V, Sperduti I, Tomao L, Forastiere E. Perioperative changes in pro and anticoagulant factors in prostate cancer patients undergoing laparoscopic and robotic radical prostatectomy with different anaesthetic techniques. J Exp Clin Cancer Res. 2014 Aug 17;33(1):63. doi: 10.1186/s13046-014-0063-z. PMID 25129475